CLINICAL TRIAL: NCT01348256
Title: Randomized Phase II Study With Dendritic Cell Immunotherapy in Patients With Resected Hepatic Metastasis of Colorectal Carcinoma
Brief Title: Study With Dendritic Cell Immunotherapy in Resected Hepatic Metastasis of Colorectal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-2009-01; 2008-007795-23 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Carcinoma; Hepatic Metastasis
Keywords: colorectal carcinoma; resectable hepatic metastasis; adjuvant treatment; dendritic cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): Observation after standard treatment
- Dendritic cells vaccine (Experimental): Adjuvant treatment with dendritic cells vaccine after standard treatment
  Interventions: Drug: Dendritic cells vaccine

INTERVENTIONS:
Drug: Dendritic cells vaccine — Vaccination with autologous dendritic cells loaded with autologous tumor antigens
  Arms: Dendritic cells vaccine

SUMMARY:
In this randomized multicentric phase II study, patients with colorectal carcinoma with resectable hepatic metastasis will be randomized to treatment with dendritic cells or to observation, following conventional treatment with surgery and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Confirmed diagnosis of colorectal cancer with hepatic metastasis, amenable for surgical treatment.
3. Capacity of understanding and signing the informed consent and to undergo the study procedures
4. Availability of tumor tissue, for maturing dendritic cells
5. Adequate renal, hepatic and bone marrow function

Exclusion Criteria:

1. Clinically relevant diseases or infections.
2. Concurrent participation in other clinical trial or administration or other antitumoral treatment
3. Concurrent cancer, with the exceptions allowed by the principal investigator (PI).
4. Pregnant or breast feeding women
5. Immunosuppressant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2010-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival | Progression free survival at 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Melero, MDPhD, Study Chair — University of Navarra
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre

REFERENCES:
- [Derived] Rodriguez J, Castanon E, Perez-Gracia JL, Rodriguez I, Viudez A, Alfaro C, Onate C, Perez G, Rotellar F, Inoges S, Lopez-Diaz de Cerio A, Resano L, Ponz-Sarvise M, Rodriguez-Ruiz ME, Chopitea A, Vera R, Melero I. A randomized phase II clinical trial of dendritic cell vaccination following complete resection of colon cancer liver metastasis. J Immunother Cancer. 2018 Sep 29;6(1):96. doi: 10.1186/s40425-018-0405-z. PMID 30268156